CLINICAL TRIAL: NCT00652223
Title: Safety, Immunogenicity and Clinical Efficacy of an Allergen Vaccine (AllQbG10) in Subjects With Allergic Rhino-Conjunctivitis and Asthma Due to House Dust Mite Allergy
Brief Title: Effect of an Allergen Vaccine in Patients With Allergic Rhino-Conjunctivitis and Asthma Due to House Dust Mite Allergy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYT005-AllQbG10 01
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Perennial Allergic Rhinoconjunctivitis; Allergic Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: CYT005-AllQbG10

INTERVENTIONS:
Biological: CYT005-AllQbG10 — Immunomodulator CYT003-QbG10 in combination with commercial house dust mite extract as used for routine SIT

SUMMARY:
The purpose of the study is to test the safety, tolerability, immunogenicity and clinical efficacy of the combination treatment AllQbG10 in patients with rhino-conjunctivitis and asthma due to house dust mite allergy in a single-center, open-label setting.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate perennial allergic rhinoconjunctivitis due to sensitization against house dust mites
* Mild asthma
* Females only if non-reproductive or agree to practice an effective and accepted method of contraception

Exclusion Criteria:

* Relevant cardiovascular, renal, pulmonary or endocrine disease
* History of autoimmune disease
* Severe allergies
* History of active infectious disease
* Current diagnosis or history of malignancy
* Relevant neurological or psychiatric disorder
* Pregnancy or lactation
* History of alcohol abuse or other recreational drugs
* Use of an investigational drug within three month before enrolment
* Blood donation within 30 days before enrolment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-03; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Mueller, MD, Study Director — Cytos Biotechnology AG
Locations (1):
- University Hospital Zurich, Department of Dermatology, Zurich, Canton of Zurich, Switzerland